CLINICAL TRIAL: NCT04182425
Title: Real-life Study to Assess the Incidence of Allergic Manifestations and Infectious Episodes in Healthy Term Infants at Risk of Dysbiosis During the First Year of Life
Brief Title: Incidence of Allergic Manifestations and Infectious Episodes in Healthy Term Infants at Risk for Dysbiosis
Acronym: SOPRANO
Status: Completed | Type: Observational
Sponsor: Bledina (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A01725-52
Record Dates: First submitted 2019-11-18; First posted 2019-12-02 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Dermatitis, Allergic Contact; Infectious Diseases
MeSH Terms: conditions — Dermatitis, Allergic Contact; Communicable Diseases | interventions — Infant Formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Infant formula — Healthy full-term infants fed on an infant formula marketed on the French market

SUMMARY:
This study will evaluate the incidence of allergic manifestations (the first of which is atopic dermatitis) and infectious diseases in children fed with an infant formula under real conditions of use.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the cumulative incidence of atopic dermatitis in healthy infants at risk for dysbiosis at 12 months of age and to identify factors associated with the presence of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* full-term infant (gestational age ≥ 37 and ≤ 42 weeks) in good health;
* Having at least one risk factor for dysbiosis, including:

  * birth by caesarean section,
  * Antibiotic exposure between birth and inclusion or in utero (mother who received antibiotics) during the last trimester of pregnancy, or per-partum (mother who received antibiotics during childbirth),
  * a family history of allergy confirmed by a doctor in a family member, affecting at least one of the two parents or siblings (asthma, atopic dermatitis, eczema, allergic rhinitis, proven food allergy);
* Aged at most 5 weeks;
* Having a weight in the reference values for gestational age and sex (between the 10th and the 90th percentiles according to the growth curves in force);
* Already consuming an infant formula (with or without associated breast milk), or whose mother wishes to introduce an infant formula at the end of this consultation to switch to mixed breastfeeding or to start weaning;
* Authorization of a parent (or both) or legal representative of the child to collect personal information about their child and family.

Exclusion Criteria:

* Premature infants or low birth weight (< 2500g);
* Infant allergic to cow's milk protein;
* Infants with severe congenital anomalies that may impact growth (cystic fibrosis, bronchopulmonary dysplasia, tracheomalacia, tracheoesophageal fistula, congenital heart defects ...);
* Infants with chronic disease or severe neonatal pathology, or a pathology predisposing to infections (HIV, hepatitis B or C, autoimmune diabetes, immune deficiency, respiratory distress, sepsis, intraventricular hemorrhage, severe neonatal hepatitis, necrotizing enterocolitis, hypertension persistent pulmonary ...), or renal or hepatic pathology;
* Inability of the parent or legal representative to understand the protocol of the study, or doubts of the physician on the ability or willingness to comply with the protocol.

Max Age: 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants up to 1 month + 1 week, in good health, at risk of dysbiosis
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis in the infants included in the study | 12 months
  Number of episodes of dermatitis reported during the 12 months of follow-up, and objectified by a SCORAD score > 0.

SECONDARY OUTCOMES:
Atopic dermatitis | 3, 6 and 12 months
  Cumulative incidence of episodes of moderate atopic dermatitis (SCORAD score of 25 to 50) or severe episodes (SCORAD score> 50)
Gastrointestinal tolerance | 3, 6 and 12 months
  * Frequency, consistency, color and quantity of stool (Amsterdam scale),
  * Frequency and intensity of regurgitations (adapted score of Vandenplas),
  * Frequency and intensity of gas / bloating, colic, unexplained crying
Height | 3, 6 and 12 months
  Growth in term of height
Weight | 3, 6 and 12 months
  Growth in term of weight
Cranial perimeter | 3, 6 and 12 months
  Growth in terme of cranial perimeter
Observance | 3, 6 and 12 months
  % of children who consumed the formula prescribed by the doctor at the previous visit
Consumption | 3, 6 and 12 months
  Number of days of consumption during the previous period.
Satisfaction with Likert scale | 3, 6 and 12 months
  5-level Likert scale filled in by the doctor and by parents
Cumulative incidence of allergic manifestations | 3, 6 and 12 months
  Cumulative number since the inclusion of episodes of:
  * atopic dermatitis,
  * eczema,
  * wheezing,
  * allergic rhinitis
Cumulative incidence of infections | 3, 6 and 12 months
  Cumulative number since the inclusion of episodes of:
  * Infection of the upper respiratory tract,
  * Infection of the lower respiratory tract,
  * Gastrointestinal infections,
  * pyelonephritis,

CONTACTS AND LOCATIONS:
Overall Officials: Florence MD CAMPEOTTO, Study Chair — Scientific Committee; Hugues MD PILOQUET, Study Chair — Scientific Committee; Alexis MD MOSCA, Study Chair — Scientific Committee; Olivier MD GOULET, Study Chair — Scientific Committee; Marie-José MD BUTEL, Study Chair — Scientific Committee; Anne-Judith MD WALIGORA, Study Chair — Scientific Committee
Locations (1):
- Medical Office, Taverny, France